CLINICAL TRIAL: NCT07387159
Title: Prospective, Interventional, Single-center Study to Evaluate the Influence of MiYOSMART iQ Spectacle Lenses With DIMS and Triple Enhanced Design Technology on Refraction Dynamics, Biometric Parameters, Peripheral Refraction and Contrast Sensitivity in Children With Myopia
Brief Title: Effect of MiYOSMART iQ Spectacle Lenses on Myopia Progression in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoya Lens Rus LLC (Industry)
Collaborators: Helmholtz National Medical Research Center of Eye Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIYOSMART-iQ-OFT-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Myopia, Child Myopia Progression
Keywords: myopia control, spectacle lenses, peripheral defocus, DIMS, MiYOSMART
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiYOSMART iQ intervention group (Experimental): DIMS with Triple Enhanced Design technology
  Interventions: Device: MiYOSMART iQ spectacle lenses
- Historical control group (No Intervention): Retrospective data from patients with single-vision spectacle correction

INTERVENTIONS:
Device: MiYOSMART iQ spectacle lenses — MiYOSMART iQ are single-vision spectacle lenses made of polycarbonate (refractive index 1.59) featuring Defocus Incorporated Multiple Segments (DIMS) technology with Triple Enhanced Design (TED). The lens contains a central optical zone for clear distance vision, surrounded by multiple, uniformly distributed micro-lens segments (diameter: ~1.00 mm) that create a consistent myopic defocus signal of +4.50 D across the peripheral retina. This specific optical design aims to slow axial elongation in progressing myopia. The intervention involves full-time wear of spectacles with these lenses. The device is CE-marked and has Russian registration certificate No. ФСЗ 2012/11555 dated December 5, 2024
  Arms: MiYOSMART iQ intervention group

SUMMARY:
This prospective, single-center study aims to evaluate the efficacy and safety of MiYOSMART iQ spectacle lenses with DIMS (Defocus Incorporated Multiple Segments) and Triple Enhanced Design (TED) technology in slowing myopia progression in children aged 8-11 years.

35 children with myopia (spherical equivalent -0.5 to -6.0 D) will be prescribed MiYOSMART iQ lenses and followed for 6 months. The study will compare changes in spherical equivalent refraction and axial length against a historical control group (n=35) using ANCOVA. Secondary outcomes include measurements of peripheral refraction and contrast sensitivity at the first prescription.

The study hypothesis is that wearing MiYOSMART iQ lenses for 6 months significantly slows myopia progression compared to single-vision spectacle correction.

DETAILED DESCRIPTION:
Introduction and Scientific Rationale Progressive myopia in children is a global public health problem associated with an increased risk of ocular pathology in adulthood. Existing myopia control methods demonstrate efficacy, but there is a need for additional non-pharmacological, non-invasive approaches with a high safety profile and patient acceptability.

MiYOSMART iQ spectacle lenses with DIMS and Triple Enhanced Design (TED) technology represent a modern method of optical myopia control, based on the concept of peripheral myopic defocus.

The efficacy of MiYOSMART lenses has been proven in a number of studies, primarily in Asian populations. However, some physiological aspects of their effect, especially in Caucasian populations and in real-world clinical practice, require further study:

Insufficient data on the precise pattern of induced peripheral defocus when using open-field instruments.

Lack of studies on the effect of defocus segments on contrast sensitivity.

Need for evaluation of key parameter dynamics (refraction, AL) in Russian children.

Scientific Hypothesis: Wearing MiYOSMART iQ spectacles for 6 months leads to a statistically significant slowing of myopia progression (by SE and AL) compared to historical control and causes characteristic, measurable changes in peripheral refraction and contrast sensitivity parameters, detectable at first prescription.

Study Objectives and Endpoints

- Primary Objective To evaluate the effect of MiYOSMART iQ spectacle lenses on myopia progression after 6 months of wear compared to a historical control group.

Primary Endpoints:

Change in Spherical Equivalent of refraction (SE, D) under cycloplegia (Visit 3 - Visit 1).

Change in Axial Length (AL, mm) (Visit 3 - Visit 1).

- Secondary Objectives

To characterize the state of the visual system at the first prescription of MiYOSMART iQ lens correction.

Endpoint 1: Peripheral refraction (D) indicators at various retinal points, measured with an open-field autorefractometer without correction and with new spectacles at Visit 2.

Endpoint 2: Spatial contrast sensitivity (log units) indicators for various spatial frequencies, measured with the "Mesotest" device in a trial frame and with new spectacles at Visit 2.

To assess the tolerability and safety of MiYOSMART iQ lens correction over 6 months.

Endpoint: Frequency, nature, and severity of all recorded Adverse Events (AEs) and Device Deficiencies (DDs).

Study Design and Methodology

* Overall Design. Prospective, interventional, single-center study with a historical control group. Responsibility for conduct and scientific supervision rests with the Principal Investigator - Elena P. Tarutta.
* Visits and Procedures. The overall schedule is presented below.

Visit 1 (Day 0, Baseline): Informed Consent, Medical History; Visual Acuity (uncorrected, with habitual and optimal correction); Autorefractometry (narrow/wide pupil); Biometry (Axial Length); Binocular Vision, Phoria, AC/A Ratio; Choroidal Thickness Measurement; Recording of Adverse Events/Device Deficiencies.

Visit 2 (within 3±1 weeks after V1): Visual Acuity with new MiYOSMART iQ spectacles; Contrast Sensitivity (Mesotest) in trial frame and new spectacles; Peripheral Refraction without correction and with new spectacles; Dispensing of MiYOSMART iQ spectacles; Recording of Adverse Events/Device Deficiencies.

Visit 3 (Month 6±1 after V1): Visual Acuity with MiYOSMART iQ spectacles; Autorefractometry; Biometry (Axial Length); Binocular Vision, Phoria, AC/A Ratio; Choroidal Thickness Measurement; Recording of Adverse Events/Device Deficiencies.

- Historical Control Group. Formed retrospectively from the research center's database. Includes patients who met the current study criteria and used single-vision spectacle correction for at least 6 months. Groups will be matched by age (±1 year) and baseline SE (±0.5 D).

ELIGIBILITY:
Inclusion Criteria:

* Age 8-11 years (inclusive)
* Myopia: spherical equivalent -0.5 to -6.0 D under cycloplegia
* No previous myopia control treatment
* Orthophoria, presence of binocular vision

Exclusion Criteria:

* Corrected visual acuity < 0.8 (decimal)
* Anisometropia > 2.0 D
* Strabismus history or presence
* Previous refractive or intraocular surgery

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | Baseline to 6 months
  Change in axial length, measured in millimeters (mm)
Change in Spherical Equivalent Refraction | Baseline to 6 months
  Change in cycloplegic spherical equivalent refraction, measured in diopters (D)

SECONDARY OUTCOMES:
Peripheral Refraction | At first prescription (Visit 2, within 3±1 weeks after baseline)
  Peripheral refraction values at various retinal points (e.g., 20° and 30° nasally, temporally, superiorly, inferiorly), measured in diopters (D) with an open-field autorefractometer, without correction and with new MiYOSMART iQ spectacles
Contrast Sensitivity | At first prescription (Visit 2, within 3±1 weeks after baseline)
  Spatial contrast sensitivity (log units) for various spatial frequencies, measured with the "Mesotest" device in a trial frame and with new MiYOSMART iQ spectacles
Safety - Incidence of Adverse Events | Throughout the study period, up to 6 months
  Frequency, nature, and severity of all recorded Adverse Events (AEs) and Device Deficiencies (DDs) related to the use of MiYOSMART iQ spectacles.

CONTACTS AND LOCATIONS:
Locations (1):
- Helmholtz National Medical Research Center of Eye Diseases, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) underlying the results reported in this study will not be publicly shared due to sponsor's data management policies, restrictions in the study contract, and confidentiality considerations regarding pediatric patient data.